CLINICAL TRIAL: NCT04232306
Title: The Effect of Liposomal Bupivacaine Plus Bupivacaine Versus Bupivacaine Alone on Postoperative Opioid Use After Elective Cesarean Delivery: a Randomized Control Trial
Brief Title: Liposomal Bupivacaine + Bupivacaine vs. Bupivacaine Alone on Opioid Use After Elective c/Section
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of resources to continue.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00081325; Pro00022425 (Other: Atrium)
Record Dates: First submitted 2019-11-19; First posted 2020-01-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain; Cesarean Section
Keywords: Postoperative analgesia; Postoperative opioid use
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, active-controlled trial
Who Masked: Participant
Masking Description: Patients will be blinded to treatment arm to which patients are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine + Bupivacaine HCL (Experimental): Liposomal bupivacaine + bupivacaine HCl surgical-site incision infiltration following spinal anesthesia
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine HCl
- Bupivacaine HCl surgical-site incision infiltration (Active Comparator): Bupivacaine HCl surgical-site incision infiltration following spinal anesthesia
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Liposomal bupivacaine — Bupivacaine liposome injectable suspension
  Other Names: Exparel
  Arms: Liposomal Bupivacaine + Bupivacaine HCL
Drug: Bupivacaine HCl — Bupivacaine HCl surgical-site incision infiltration
  Other Names: Bupivacaine

SUMMARY:
The purpose of this study is to compare the effectiveness of local wound infiltration of EXPAREL® (liposomal bupivacaine) with bupivacaine HCl compared to active control with bupivacaine HCl alone following elective primary or repeat cesarean delivery with spinal anesthesia.

DETAILED DESCRIPTION:
Pain in the postpartum period is an important concern of new mothers. With over one-third of deliveries ending in cesarean section, effective postoperative pain control is essential in the care of postpartum patients.1 Improved pain control in the postpartum period after cesarean delivery (CD) is associated with improved overall maternal health and satisfaction, decreased postpartum depression, shortened hospital stay, decreased opioid consumption, and decreased healthcare costs, as well as possible facilitation of early contact of mothers with their infants.2 Pain control is of great concern to women during and after cesarean delivery.3 Pain relief and patient satisfaction are inadequate in many cases. Pain may be severe, last at least 48-72 hours, and may impair early postoperative recovery.

Opioids are primarily used in the post-operative period. Although opioids are safe to use in breastfeeding mothers, they are not without unwanted side effects.4 Local anesthetics and parenteral NSAIDs are also beneficial adjuncts to regional or general anesthesia after CD by reducing opioid consumption and improving pain relief.5 In addition, field block with wound infiltration with local anesthetic is an effective and safe adjunct for pain control. Previous studies have shown improved postoperative pain control with TAP (transversus abdominis plane) blocks with bupivacaine in hysterectomy patients.4 Another study has looked at the effects of bupivacaine-soaked spongostan placed in cesarean wounds.2 EXPAREL®® (Parsippany, NJ: Pacira Pharmaceuticals, Inc) is a liposomal form of bupivacaine. Its mechanism of action is by DepoFoam® technology, in which microscopic, polyhedral molecules that contain aqueous chambers with liposomal bupivacaine that are slowly released over hours to days with erosion and rearrangement of lipid membranes.6 The slow release of local anesthetic extends its pharmacologic effect and provides longer postsurgical pain control for up to 72 hours.6 This method of delivery of local anesthetic has the potential to decrease postoperative opioid consumption.7 EXPAREL® is an FDA-approved medication for the general use of postoperative surgical site pain control. Paracervical block is the only obstetric contraindication to EXPAREL® use. The purpose of this study is to compare the effectiveness of local wound infiltration of EXPAREL® (liposomal bupivacaine) with bupivacaine HCl compared to active control with bupivacaine HCl alone following elective primary or repeat cesarean delivery with spinal anesthesia. The investigators hypothesize that narcotic use during postoperative hospitalization will be decreased using liposomal bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age and older at screening
* Subjects at 37 completed weeks of gestation or greater undergoing elective primary or repeat cesarean delivery (CD)
* Pfannenstiel incision
* Regional spinal anesthesia
* ASA classification I, II, or III
* Able to give informed consent
* English- or Spanish-speaking

Exclusion Criteria:

* ASA classification IV
* Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (eg, amide-type local anesthetics, opioids, bupivacaine, NSAIDs, spinal anesthesia).
* Potential drug interaction(s) with bupivacaine
* Severe renal or hepatic dysfunction manifest as serum creatinine level >2 mg/dL, blood urea nitrogen level >50 mg/dL , serum aspartate aminotransferase level >3 times the upper limit of normal, or serum alanine aminotransferase level >3 times the ULN.
* Any clinically significant maternal or fetal event or condition arising during surgery (eg, excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course. In this situation, the subject would be ineligible to receive study drug and withdrawn from the study.
* Chronic pain disorder manifest as a concurrent, painful, physical condition that may require long-term, consistent use of opioids postoperatively for pain that is not strictly related to the surgery and may confound postsurgical assessments.
* History of, suspected, or known addiction or abuse of illicit drug(s) or prescription medication(s) within the past 2 years.
* Planned concurrent surgical procedure except for salpingo-oophorectomy or tubal ligation.
* Subject at increased risk for bleeding or coagulation disorder (defined as platelet count less than 80,000/mm3 or international normalized ratio[INR] greater than 1.5).
* Pregnancy body mass index >50 kg/m2 or otherwise not anatomically appropriate to undergo local incision infiltration.
* Conversion of spinal anesthesia to general anesthesia due to incomplete neuraxial block and unsatisfactory surgical anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility based on gender female
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Amount of total opioid MME (milligram morphine equivalents) consumed at 24, 48 and 72hrs post-op | 72 hours
  3.1 To compare total opioid consumption through 72-hours following EXPAREL® + bupivacaine HCl surgical-site infiltration versus bupivacaine HCl alone at elective primary or repeat cesarean delivery after spinal anesthesia. 3.2 Primary outcome of this study is total opioid consumption measured in milligram morphine equivalents (MME) at 24-, 48- and 72-hours postoperatively and total MME for duration of hospital admission.

SECONDARY OUTCOMES:
time to initial rescue analgesia administration | 24 hours
  Time in hours and minutes
Numeric Pain Rating Score at 72 hours Postoperative | 72 hours
  postoperative pain assessment with NRS (Numeric Pain Rating Score). NRS score is comprised of 4 pain questions with the patient rating each one on a scale of 0(no pain) to 10(worst pain imaginable). Lower scores are favorable.
Overall Benefit of Analgesia Score at 72 hours Postoperative | 72 hours
  postoperative pain assessment with OBAS (Overall Benefit of Analgesia Score). The OBAS is comprised of 7 questions each being scored by the patient from 0(minimal pain) to 4(maximum imaginable pain). Each question is then added up to total the overall benefit of analgesia score. Lower scores are favorable.
Length of hospital stay | 72 hours
  measured in days and hours
Initiation of breastfeeding | 72 hours
  yes/no and time to initiation as measured in days and hours
Postpartum depression scores | 72 hours
  PHQ-9 postpartum depression scores. Possible range is 0-27. Lower scores mean less depression.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Boardman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared